CLINICAL TRIAL: NCT06417918
Title: A Formative Study to Develop Culturally Valid Psychosocial Assessment Tools and Interventions to Promote Family Well-Being in Kenya - Part II
Brief Title: An Evaluation of a Family Counseling Intervention ("Tuko Pamoja") in Kenya
Acronym: C0058 (4C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Moi University (Other)
Responsible Party: Principal Investigator, Eve Puffer, Director, Duke Center for Global Mental Health; Associate Professor, Psychology and Neuroscience and Global Health, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0210 (4C)
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Issue; Family Relations; Family Conflict; Child Mental Disorder; Adolescent - Emotional Problem; Adolescent Problem Behavior; Child Behavior; Child Abuse; Marital Conflict; Domestic Violence; Parent-Child Relations; Parenting
MeSH Terms: conditions — Neurodevelopmental Disorders; Child Behavior

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Tuko Pamoja (Experimental): The intervention, Tuko Pamoja, is in-home family counseling delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices including family systems and solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. The content and structure has been adapted based on formative research in this context. Tuko Pamoja is manualized and includes a tablet-based manual material and video content to support psychoeducation components and data collection.
  Interventions: Behavioral: Tuko Pamoja, "We are Together" in Kiswahili
- Control (No Intervention): Waitlist control (will receive the in-home counseling after the final data collection point)

INTERVENTIONS:
Behavioral: Tuko Pamoja, "We are Together" in Kiswahili — Tuko Pamoja, "We are Together" in Kiswahili; This intervention, delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include solution-focused family therapy and cognitive behavioral strategies. It is components based, with modules delivered based on need. Tuko Pamoja includes a smart phone component to support psychoeducation components and data collection. The content and structure has been adapted in both content and implementation model based on formative research in this context.
  Arms: Intervention: Tuko Pamoja

SUMMARY:
The purpose of this study is to evaluate a family counseling intervention, entitled "Tuko Pamoja" (Translation "We are Together" in Kiswahili). The intervention, delivered by lay counselors and through existing community social structures, is expected to improve family functioning and individual mental health among members. The sample includes families with a child or adolescent (ages 8-17) experiencing problems in family functioning.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a family counseling intervention, entitled "Tuko Pamoja" (Translation "We are Together" in Kiswahili), using a pilot randomized control trial design.

The intervention, delivered by lay counselors and through existing community social structures, focuses on improving family relationships and mental health with content derived from evidence-based practices; these include family systems and solution-focused family therapies and cognitive behavioral strategies. It is components based, with modules delivered based on need. The content and structure has been adapted in both content and implementation model based on formative research in this context. Primary hypotheses include achieving improvements in outcomes related to:

1. Family functioning, including elements such as communication, emotional closeness, structure and organization, and satisfaction for the overall family; this also includes indicators of functioning at dyadic levels (i.e., parent-child and couples functioning)
2. Mental health of both children and caregivers.

The investigators also hypothesize feasibility and acceptability, including high fidelity and adequate clinical competency by the non-specialist counselors, based on a previous evaluation of the program.

The study will follow a randomized controlled design with a target sample size of 60 families, including up to 2 caregivers per family (who hold primary responsibility for the child whether biological or non-biological) and a target child identified either through caregiver-report of the child about whom they are most concerned or randomly, if there is no child with particular concerns. Families will be recruited in two rounds of 30 families due to logistical limitations of enrolling all 60 at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Family with self-reported elevated distress (e.g., high levels of conflict) that also has a child/adolescent (ages 8-17) with caregiver-reported emotional or behavioral concerns

Exclusion Criteria:

* Families without reported distress and/or without reported adolescent distress.
* Families with children older than 17 or younger than 8 years of age.
* Families in which primary caregivers or children are living too far outside of the community to participate in treatment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Family Functioning (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  30 self-report items developed for the local context based on formative research (Family Togetherness Scale, FTS). Responses are endorsed on a 10-point scale and refer to the past month. One composite score is calculated (range: 0 - 30); higher scores represent more family distress.
Parent-Child Communication (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  20 self-report items from the Parent-Adolescent Communication Scale (PACS). Each include caregiver and child/adolescent report versions. Participants are asked to respond based on the past month. Children report on each caregiver separately. One composite score is calculated (range: 0 - 60); higher scores represent better parent-child communication.
Parent-Child Relationship Quality (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  20 self-report items from the Parent Adolescent Relationship Questionnaire (PARQ) Warmth Subscale. One composite score is calculated (range: 0 - 60); higher scores represent better parent-child relationship quality.
Harsh Parenting (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  15 self-report items from the Parent Adolescent Relationship Questionnaire (PARQ) Hostility/Aggression Subscale. One composite score is calculated (range: 0 - 45); higher scores represent more harsh parenting characteristics.
Couples Relationship Quality (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  13 self-report items from the Dyadic Adjustment Scale (DAS) Cohesion and Satisfaction subscales and 9 locally-developed items. One composite score is calculated (range: 22 - 132); higher scores represent better couples relationship quality.
Child Mental Health (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  20 self-report items from the Child Behavior Checklist (CBCL) and 6 locally-developed items. One composite score is calculated (range: 20 - 60); higher scores represent worse child mental health.
Child Mental Health (Child Report) | Baseline, 1 month, and 3 month post-intervention
  19 self-report items from the Youth Self-Report (YSR) and 7 locally-developed items. One composite score is calculated (range: 0 - 52); higher scores represent worse child mental health.
Caregiver Mental Health (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  9 self-report items from the Patient Health Questionnaire (PHQ-9), 14 self-report items from the General Health Questionnaire (GHQ), and 6 locally-developed items. One composite score is calculated (range: 0 - 87); higher scores represent worse caregiver mental health.

SECONDARY OUTCOMES:
Physical Maltreatment (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  2 items from the Multiple Indicator Cluster Survey (MICS) and 2 items from the Discipline Interview. One composite score is calculated (range: 0 - 12); higher scores represent more physical maltreatment.
Couples Violence (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  3 locally-developed items. One composite score is calculated (range: 0 - 12); higher scores represent more couples violence.
Child Belongingness in Family (Child Report) | Baseline, 1 month, and 3 month post-intervention
  5 locally-developed items. One composite score is calculated (range: 0 - 10); higher scores represent more child belongingness in the family.
Child Hope (Child Report) | Baseline, 1 month, and 3 month post-intervention
  6 self-report items from the Children's Hope Scale. One composite score is calculated (range: 6 - 36); higher scores represent higher hope levels.
Child Prosocial Behavior (Caregiver and Child Report) | Baseline, 1 month, and 3 month post-intervention
  6 locally-developed items. One composite score is calculated (range: 0 - 12); higher scores represent more prosocial behaviors.
Caregiver Hope (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  12 self-report items from the Children's Hope Scale. One composite score is calculated (range: 6 - 48); higher scores represent higher hope levels.
Social Support (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  28 self-report items from the Inventory of Socially Supportive Behaviors (ISSB), 12 self-report items from the Multidimensional Scale of Perceived Social Support (MSPSS), and 7 locally-developed items. One composite score is calculated (range: 29 - 147); higher scores represent more social support.
Child Well-being (Child Report) | Baseline, 1 month, and 3 month post-intervention
  7 self-report items from the Short Warwick Edinburgh Well-being Scale. One composite score is calculated (range: 7 - 35); higher scores represent better child well-being.
Adult Well-being (Adult Report) | Baseline, 1 month, and 3 month post-intervention
  7 self-report items from the Short Warwick Edinburgh Well-being Scale. One composite score is calculated (range: 7 - 35); higher scores represent better adult well-being.
Caregiver Coping (Caregiver Report) | Baseline, 1 month, and 3 month post-intervention
  28 self-report items from the Brief-COPE. One composite score is calculated (range: 28 - 112); higher scores represent better coping skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No